CLINICAL TRIAL: NCT02916004
Title: Responsiveness to Noxious Stimuli in Ventilated Intensive Care Unit (ICU) Patients With Propofol / Remifentanil Sedation Protocol by Using the Nociception Flexion Reflex (RIII Reflex) and the Pupillary Dilatation Reflex.
Brief Title: The Use of Nociception Flexion Reflex and Pupillary Dilatation Reflex in ICU Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Davina Wildemeersch, MD, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16/33/334
Record Dates: First submitted 2016-09-15; First posted 2016-09-27 (Estimated); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Critical Illness
Keywords: Analgesia; Pain measurement; Nociception; Electromyography; Electrical stimulation; Pupillometry; Critical care; Sedation
MeSH Terms: conditions — Critical Illness; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Measurement of NFR and PDR (Other): Diagnostic intervention: excite NFR and PDR in comparison to behavior pain scale (BPS)
  Interventions: Device: Measurement of NFR and PDR

INTERVENTIONS:
Device: Measurement of NFR and PDR — Feasibility testing of NFR and PDR in sedated, ventilated patients. Comparison of NFR and PDR with standard routine care of pain assessment

SUMMARY:
The aim of the study was to describe the feasibility of the nociception flexion reflex and the pupillary dilatation reflex as objective pain assessment tools in the Intensive Care Unit (ICU). Furthermore to describe the relationship between the responses and the standard of care pain evaluation in the critically ill sedated patients.

Patients were under propofol / remifentanil or propofol / sufentanil sedation protocol during measurements in a stair-case increasing intensity model of standardized stimulations. (Stimulation intensity are similar to the stimulations of neuromuscular blocking agents monitoring.)

DETAILED DESCRIPTION:
Pupillary dilatation reflex: tetanic stimulations at the nervus medianus were performed starting form 10 milliamperes (mA) up to 60mA. Pupillary diameter was measured before, during and after stimulation.

Nociception flexion reflex: tetanic stimulations at the nervus suralis were performed starting form 0.5mA in increasing steps via an automated RIII (NFR) threshold tracking model.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Critically ill with necessity to mechanic ventilation
* Hospitalized at the ICU of our institution
* Started sedation protocol (propofol/remifentanil or propofol/sufentanil)
* Approved informed consent by family member or relative.

Exclusion Criteria:

* Known eye deformity or extented ophthalmologic surgery in history
* Severe traumatic brain injury of fulminant stroke
* Known (poly)neuropathy of complicated diabetes
* Need for continuously curarization
* Hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09-26 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-07-14 (Actual)

PRIMARY OUTCOMES:
Test the feasibility of a objective pain evaluation tool; the nociception flexion reflex (NFR) | 10 seconds after nociceptive stimulation
Test the feasibility of a objective pain evaluation tool; the pupillary dilatation reflex (PDR) | 10 seconds after nociceptive stimulation

SECONDARY OUTCOMES:
Comparison NFR and the standard of care pain assessment (behavior pain scale) | In period of routine two hourly check up by nurse
  Routine assessment of pain by attending nurse
Comparison PDR and the standard of care pain assessment (behavior pain scale) | In period of routine two hourly check up by nurse
  Routine assessment of pain by attending nurse

CONTACTS AND LOCATIONS:
Overall Officials: Davina Wildemeersch, MD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University hospital Antwerp, Edegem, Antwerpen, Belgium